CLINICAL TRIAL: NCT06130631
Title: Retrospective Study on Predictors of Steroid Response in Childhood Nephrotic Syndrome at Assiut University Children Hospital
Brief Title: Predictors of Steroid Response in Childhood Nephrotic Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maha Radwan (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Maha Radwan, 71515, Assuit, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Steroid in nephrotic syndrome
Record Dates: First submitted 2023-11-04; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Nephrotic Syndrome in Children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective study of predictors of steroid response in childhood nephrotic syndrom

DETAILED DESCRIPTION:
Nephrotic syndrome is the most common glomerular disease affecting children worldwide ,Nephrotic syndrome is the combination of nephrotic-range proteinuria with a low serum albumin level and edema. Nephrotic-range proteinuria is the loss of 3 grams or more per day of protein into the urine or, on a single spot urine collection, the presence of 2 g of protein per gram of urine creatinine. Minimal change disease (MCD) or minimal change glomerulonephritis and focal segmental glomerulosclerosis (FSGS) are the two major causes of nephrotic syndrome in children and young adults, Idiopathic, hereditary, and secondary forms are due to underlying increased protein leakiness across the glomerular capillary wall, as a result of immune and non-immune insults affecting the podocyte.

The incidence worldwide varies widely between 1.2 and 16.9 cases per 100,000 children with the highest incidence observed on the Indian subcontinent compared to 2-3 cases per 100,000 children in most other regions . Males appear to be more affected than females at a ratio of 2:1 at a younger age, but this predominance fails to persist in adolescence.

treatment of nephrotic syndrome:- Corticosteroids have been used to treat childhood nephrotic syndrome since 1950 when large doses of adrenocorticotrophic hormone (ACTH) and cortisone given for two to three weeks were found to induce diuresis with loss of oedema and proteinuria. The response to treatment with steroids has been shown to vary by ethnicity, likely due to environmental and genetic factors. Corticosteroid usage has reduced the mortality rate in childhood nephrotic syndrome to around 3%, with infection remaining the most important cause of death. Of children who present with their first episode of nephrotic syndrome, approximately 80% will achieve remission with corticosteroid Prednisolone is the mainstay treatment, whose response is often presumed to determine the long-term risk of disease progression and is a better prognostic indicator . Although patients with steroid-sensitive nephrotic syndrome generally have good outcomes, more than half will have a frequently relapsing course and steroid dependence. Up to 95% of patients with minimal change nephrotic syndrome (MCNS) attain complete remission after an 8-week course of high dose steroids there are some factors affecting response to treatment with the steroids such as age of onset (the older the age of onset the better the response) ,gender (the females respond more to treatment) and type of nephrotic syndrome( minimal change glomerulonephritis responds more than focal segmental glomerulosclerosis to steroids ).

ELIGIBILITY:
Inclusion Criteria:

* all children from 1 year to 18 years treated with steroid for nephrotic syndrom

Exclusion Criteria:

* children with other kideny disease Children less than 1 year old Children with secondary nephrotic syndrom

Ages: 12 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Gender Based: Yes — All children from 1 year to 18 years
Study Population: All patient diagnosed with nephrotic syndrom on steroid treatment for 3 years
Sampling Method: Non-Probability Sample
Enrollment: 79 (Estimated)
Dates: Start 2023-12-03 (Estimated); Primary Completion 2024-12-21 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Predictors of steroid response in childhood nephrotic syndrom | 2year
  Retrospective study of predictors of steroid response in childhood nephrotic syndrom Sach as hypertension, hematuria,raised renal chemistry in pediatric nephrology unit and outpatient outpatient nephrology clinic at assiut university children hospital

CONTACTS AND LOCATIONS:
Overall Officials: Maha Radwan Zaki, Principal Investigator — Assiut University

REFERENCES:
- [Background] Anochie I, Eke F, Okpere A. Childhood nephrotic syndrome: change in pattern and response to steroids. J Natl Med Assoc. 2006 Dec;98(12):1977-81. PMID 17225845
- [Background] Sinha A, Bagga A. Nephrotic syndrome. Indian J Pediatr. 2012 Aug;79(8):1045-55. doi: 10.1007/s12098-012-0776-y. Epub 2012 May 30. PMID 22644544